CLINICAL TRIAL: NCT07006298
Title: One-year Outcomes by Index Treatment in Elderly Patients With Acute Cholecystitis: Protocol of the International, Prospective, Observational GOLDENEYE Study
Brief Title: One-year Outcomes by Index Treatment in Elderly Patients With Acute Cholecystitis
Acronym: GOLDENEYE
Status: Recruiting | Type: Observational
Sponsor: Instituto de Investigación Sanitaria y Biomédica de Alicante (Network)
Responsible Party: Principal Investigator, Nuria Lluis Viñas, MD, PhD, Instituto de Investigación Sanitaria y Biomédica de Alicante
Other Study IDs: Goldeneye Study
Record Dates: First submitted 2025-05-14; First posted 2025-06-05 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Acute Cholecystitis
Keywords: laparoscopic cholecystectomy; Conservative Treatment; drainage; Endosonography; Propensity Score; Retrospective Studies
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Supportive care: Patients that received antibiotics only
- Cholecystectomy: Patients that undergo early or delayed cholecystectomy
- percutaneous gallbladder drainage: Patients that undergo percutaneous gallbladder drainage
- EUS-guided gallbladder drainage: Patients that undergo EUS-guided gallbladder drainage

SUMMARY:
Background: The GOLDENEYE study is an international, multicenter, prospective observational investigation designed to compare the outcomes of various management strategies for acute cholecystitis in patients aged 70 years and older. This research is driven by the increasing prevalence of gallstones and biliary tract diseases in the elderly, alongside a recognition that the burden of comorbidity in this population may necessitate tailored treatment approaches to optimize outcomes.

Patients and Methods: The primary aims of the study are to evaluate the efficacy of different treatments -supportive care, percutaneous gallbladder drainage, early or delayed cholecystectomy, and EUS-guided gallbladder drainage- on patient-centric outcomes, including one-year additional treatment modalities, hospital readmissions, outpatient encounters, quality of life, and survival rates. The study adopts a robust design incorporating propensity score matching analysis to account for the non-randomized allocation of treatment modalities, thereby minimizing selection bias and enhancing the comparability of treatment groups. Inclusion criteria are centered on patients ≥70 years diagnosed with acute cholecystitis, as per the Tokyo guidelines, while key exclusion criteria include prior episodes of cholecystitis or pancreatitis, terminal illness, and concurrent diagnosis of acute pancreatitis, cholangitis, bile duct disease, or digestive malignancy. Data collection will leverage the REDCap platform for systematic and secure data management, facilitating real-time data entry and monitoring across participating centers.

Discussion: This comprehensive approach ensures the integrity and reliability of data collected on demographics, gender, clinical outcomes, and quality of life measures. Through its innovative design and methodology, the GOLDENEYE study aims to generate evidence-based insights that will significantly influence the management of acute cholecystitis in the elderly, ultimately improving patient outcomes and healthcare practices in this growing demographic population.

ELIGIBILITY:
Inclusion Criteria:

* patients ≥70 years
* diagnosed with acute cholecystitis, as per the Tokyo guidelines

Exclusion Criteria:

* prior episodes of cholecystitis or pancreatitis
* terminal illness
* concurrent diagnosis of acute pancreatitis, cholangitis, bile duct disease, or digestive malignancy

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients ≥70 years diagnosed with acute cholecystitis, as per the Tokyo guidelines
Sampling Method: Non-Probability Sample
Enrollment: 376 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2027-05-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
1 year additional procedures, hospital readmissions or outpatient visits | 1 year
  Percentage of patients requiring any additional procedure, hospital readmission or outpatient visit during the first year.

SECONDARY OUTCOMES:
1-year health-related quality of life | 1 year
  The EQ-5D-5L questionnaire is used to assess quality of life in elderly individuals. It encompasses five key dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is evaluated across five severity levels. Level 1 indicates that the patient has no problems. Level 5 indicates the worst condition. Additionally, the questionnaire has a scale. This scale is numbered from 0 to 100. A score of 100 indicates the best health possible. Zero means the worst health possible. Measurements will be obtained during the initial admission and at one, three, and twelve months.
1-year overall survival | 1 year
  Survival will be defined as the time elapsed between the date of index admission and the date of death or last follow-up. Survival curves will be constructed by the Kaplan-Meier method and compared using the log-rank test. A multivariable Cox proportional hazards regression model will be used to identify prognostic factors associated with survival. All variables that are significant at 0.10 in the univariable analysis will be entered into a multivariable model. P-values less than 0.05 will be considered statistically significant. All analyses will be performed with RStudio, version 1.2.5001 (Integrated Development for R. RStudio, Inc., Boston, MA, USA).

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Investigación Sanitaria y Biomédica de Alicante (ISABIAL), Alicante, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No
The Steering Committee and statistical advisors will have access to the final dataset. Members of the GOLDENEYE study that recruited patients may claim access to the final dataset to perform ancillary studies; the Steering Committee will study these proposals. Any data required to support the protocol can be supplied on request.

REFERENCES:
- [Derived] Lluis N, Perez-Brotons S, de Castro I, Martinez B, Aparicio JR, Zapater P, Lluis F, de-Madaria E. One-year outcomes by index treatment in older patients with acute cholecystitis. Protocol of the international, prospective, observational GOLDENEYE study. Cir Esp (Engl Ed). 2025 Dec 23:800282. doi: 10.1016/j.cireng.2025.800282. Online ahead of print. PMID 41448354
- See also: Related Info — https://ericaresearch.com/en/estudios-activos/goldeneye/